CLINICAL TRIAL: NCT06818097
Title: Efficacy Analysis of the Combined Target - Immunotherapy and XELOX Chemotherapy Regimen in the Treatment of Advanced Hepatocellular Carcinoma.
Brief Title: Efficacy of Target - Immunotherapy and XELOX Chemotherapy for Advanced HCC
Acronym: T+I+XELOX
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: TKI+PD-1+XELOX-HCC
Record Dates: First submitted 2025-01-16; First posted 2025-02-10 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-01

CONDITIONS: Advanced HCC; Systemic Therapy; Chemotherapy; Immunotherapy; Targeted Therapy; Efficacy and Safety
Keywords: TKI; XELOX; advanced HCC; PD-1 antibody
MeSH Terms: interventions — spartalizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment group: TKI+PD-1 antibody +XELOX chemotherapy
  Interventions: Drug: TKI; Drug: anti PD-1; Drug: XELOX chemotherapy

INTERVENTIONS:
Drug: TKI — Lenvatinib
Drug: anti PD-1 — Sintilimab or Camrelizumab or Tislelizumab
Drug: XELOX chemotherapy — Capecitabine and Oxaliplatin

SUMMARY:
In China, primary hepatocellular carcinoma (HCC) has high morbidity and mortality, imposing a heavy burden on the public. Surgical resection is an effective treatment, but as HCC is often latent, less than 30% of patients are suitable for surgery at first diagnosis. So systemic anti-tumor therapy is crucial for advanced HCC. Small-molecule targeted drugs like lenvatinib and sorafenib are NCCN-recommended first-line drugs for advanced HCC. The combination of targeted drugs and immune checkpoint inhibitors can prolong overall survival with good safety. The "2024 Guidelines for HCC Diagnosis and Treatment" shows that platinum-containing chemotherapy is a preferred systemic treatment for advanced HCC. However, in real-world practice, the efficacy and safety of the combination of targeted-immunotherapy and chemotherapy regimen for advanced HCC remain unclear.

DETAILED DESCRIPTION:
This study is a retrospective cohort study aimed at evaluating the efficacy and safety of TKI + PD-1 inhibitor + XELOX chemotherapy in the treatment of advanced HCC. The study included the clinical data of 68 patients with advanced HCC who could not undergo radical surgical resection and received first-line triple-drug therapy (lenvatinib as TKI + camrelizumab/ tislelizumab/ atezolizumab as PD-1 inhibitor + capecitabine and oxaliplatin as XELOX chemotherapy regimen) in the Hepatobiliary Surgery Department of Sun Yat-sen Memorial Hospital, Sun Yat-sen University from April 2022 to December 2024. Demographic information, imaging information, blood biochemistry, blood routine, alpha - fetoprotein and other information of patients were collected as baseline information. Subsequently, based on the RECIST v1.1 standard, the objective response rate (ORR) evaluated by the researchers was set as the primary endpoint, and the surgical conversion rate, overall survival (OS), progression - free survival (PFS), and the incidence of adverse events were analyzed as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Be aged 18 years or older and be diagnosed with HCC by histology, cytology, or imaging studies.
2. Have HCC with a clinical stage corresponding to Barcelona Clinic Liver Cancer (BCLC) stage C.
3. Have not undergone systemic treatment previously, and initially receive the targeted - immunotherapy combined with XELOX chemotherapy regimen (lenvatinib + Sintilimab or Camrelizumab or Tislelizumab + Capecitabine + Oxaliplatin) upon the diagnosis of HCC.
4. Have a liver function classified as Child - Pugh grade A or B.
5. Have an ECOG PS score of 0 or 1.

Exclusion Criteria:

1. Experienced rupture and bleeding of esophageal or gastric varices within the past six months.
2. Imaging findings indicate the presence of main portal vein invasion in hepatocellular carcinoma.
3. Imaging results show inferior vena cava involvement in hepatocellular carcinoma.
4. Imaging examinations reveal cardiac involvement in hepatocellular carcinoma.
5. Pregnancy and lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable liver cancer
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | from the patient's first medication use to the 6th treatment cycle, with each cycle lasting for 21 days

SECONDARY OUTCOMES:
Overall Survival | From the date of assignment to the date of death from any cause (or the date of the last follow-up if the patient was alive), with an assessment period of up to 12 months
Progression Free Survival | From the date of assignment to progression according to RECIST 1.1 or death from any cause, whichever occurred first, with an assessment period of up to 12 months.
Adverse event incidence rate | from the first cycle after treatment to 90 days after the last cycle.
Surgical conversion rate | From the date of starting treatment to the date of receiving surgical resection, assessed up to 21 days

CONTACTS AND LOCATIONS:
Locations (1):
- Sen Memorial Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No